CLINICAL TRIAL: NCT06803199
Title: Investigation of the Combined Effects of Luteinizing Hormone and Follicle-Stimulating Hormone on Metabolic Regulation in Cumulus Cells
Brief Title: Effects of LH and FSH on Metabolic Regulation in Cumulus Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH24-CT7-22
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Unrecognized Condition
MeSH Terms: interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined FSH and LH (Experimental): Participants receive combined FSH and LH during controlled ovarian stimulation in IVF cycle
  Interventions: Drug: FSH and LH
- FSH alone (Active Comparator): Participants receive combined FSH and LH during controlled ovarian stimulation in IVF cycle
  Interventions: Drug: FSH

INTERVENTIONS:
Drug: FSH and LH — In the study group, participants receive FSH and LH in IVF cycle
  Arms: combined FSH and LH
Drug: FSH — In the control group, participants receive FSH alone in IVF cycle
  Arms: FSH alone

SUMMARY:
The combined use of follicle-stimulating hormone (FSH) and luteinizing hormone (LH) has improved IVF pregnancy rates in infertile women aged 35-40, but its mechanisms remain unclear. This prospective study will examine how FSH and LH combined treatment affects cumulus cell energy metabolism. Sixty participants will be divided into two groups receiving either combined therapy or FSH alone. The study will analyze patient characteristics, infertility history, and compare mitochondrial function in cumulus cells to evaluate treatment effectiveness.

DETAILED DESCRIPTION:
The impact of combined follicle-stimulating hormone (FSH) and luteinizing hormone (LH) treatment on ovulation stimulation in older infertile women has garnered significant attention in reproductive medicine. While research indicates improved in vitro fertilization (IVF) pregnancy rates in women aged 35-40 receiving combined FSH and LH therapy compared to FSH alone, the underlying mechanisms and effectiveness remain unclear. This prospective study aims to investigate the effects of combined FSH and LH treatment on cumulus cell energy metabolism in infertile women aged 35-40 undergoing IVF treatment. The research will involve 60 participants divided into two equal groups: one receiving combined FSH and LH therapy and the other receiving FSH alone. The study will collect comprehensive data including baseline characteristics, infertility history, ovarian function parameters, and ovulation stimulation cycle outcomes. Additionally, cumulus cells will be collected from both groups to compare their mitochondrial metabolic function. Through this investigation, we seek to understand whether the combined hormone approach can enhance cumulus cell energy metabolism and improve overall ovulation stimulation outcomes in this specific age group. CopyRetryClaude can make mistakes. Please double-check responses.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-40 years
* BMI 18-30 kg/m2
* planning to undergo IVF cycles

Exclusion Criteria:

* Primary ovarian insufficiency
* history of oophorectomy
* receiving oocyte donation
* Chromosome anomaly
* Congenital uterine anomaly
* Severe intrauterine adhesion
* Malignancy
* Using hormone therapy or supplements in recent 3 months

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women planning to undergo IVF cycles
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
oxygen consumption rate of mitochodria (%) | through study completion, an average of 3 year
  to assess mitocondrial function in cumulus cells
Live birth rate (%) | through study completion, an average of 3 year
  a viable infant after 24 weeks of gestation

SECONDARY OUTCOMES:
Amount of ATP production (moles/min) of mitochodria | through study completion, an average of 3 year
  to assess mitocondrial function in cumulus cells
Clinical pregnancy rate (%) | through study completion, an average of 3 year
  the presence of a fetal heartbeat detected via transvaginal sonography at 6-7 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No